CLINICAL TRIAL: NCT05718479
Title: Reducing Stress-Sensitive Problems Among Pregnant Black Women With Childhood Adversity: A Pilot Randomized Controlled Trial of Motivational Interviewing and Mental Wellness Skills
Brief Title: Reducing Stress-Sensitive Problems Among Pregnant Black Women With Childhood Adversity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ellen Goldstein, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1175; U54MD012523 (NIH)
Record Dates: First submitted 2022-12-01; First posted 2023-02-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Maternal Psychological Distress; Perinatal Depression; Self-Regulation, Emotion
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The intervention consists of four weekly individual sessions. In Step One, participants identify ways of coping with stress and create a behavior change plan with measurable goals. An initial 1-hour semi-structured interview provides an opportunity to self-assess motivation to change a health behavior. Step Two facilitates a behavior plan assisting participants to identify a measurable goal, barriers to achieving their goal, strategies to mitigate triggers, social supports, and progress rewards. Sessions 2-4 include a 10-minute check-in to assess the status of targeted behaviors, troubleshoot potential barriers, modify the plan, and reinforce progress followed up with 20-minutes of practicing mindfulness. In Step Three, participants will learn and practice mental wellness skills (e.g., tracking, resourcing, grounding, gesturing), which can be applied to changing a behavior.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma Informed Prenatal Intervention (TPI) (Experimental): The experimental arm consists of four weekly, individual (30-60 minute) sessions via Zoom with a trained behavioral health scientist and therapist facilitating motivational interviewing focused on behavior change and mental wellness skills.
  Interventions: Behavioral: Trauma Informed Prenatal Intervention (TPI)
- Prenatal Education Topics (Active Comparator): The active comparator arm consists of four weekly, individual (30-45 minute) sessions via Zoom with a research staff member delivering prenatal education topics consisting of lecture (power point slides) and video.
  Interventions: Other: Prenatal Education Topics

INTERVENTIONS:
Behavioral: Trauma Informed Prenatal Intervention (TPI) — TPI is designed to foster behavior change and health coping by enhancing knowledge, beliefs, regulation skills and abilities. In the experimental group, a research staff member will meet with participants and help them to identify a health behavior they want to change, explore the pros and cons of making a change, create a behavior change plan, and learn several mindfulness meditation techniques. The facilitator will check-in with the participants about their behavior change plan in the subsequent sessions regarding progress made, barriers encountered, and changes in the plan and/or goal going forward. Participants will be instructed to implement an at-home mental wellness skills and provided with a tracking log to report the frequency and dose of daily/weekly practice.
  Arms: Trauma Informed Prenatal Intervention (TPI)
Other: Prenatal Education Topics — In the control group, a research staff member will provide participants with four different weekly prenatal education topics, including information on prenatal care, labor and delivery, postpartum care, and newborn care.
  Arms: Prenatal Education Topics

SUMMARY:
The goal of this clinical trial is to test the feasibility and acceptability and compare outcomes of a trauma-informed prenatal intervention (TPI) in pregnant Black women with childhood adversity. TPI participants will receive four weekly individual virtual sessions of motivational interviewing to promote self-efficacy and mental wellness skills to enhance self-awareness and self-regulation. TPI is designed to foster behavior change and health coping by enhancing knowledge, beliefs, regulation skills and abilities.

* With the assistance of a trained facilitator, participants will be guided to identify a specific goal related to the behavior they want to change.
* Behavior change goals will be individualized to create a change plan that reinforces resilience-based coping, accountability, and self-care rewards.
* Participants will learn to apply mental wellness skills to enhance regulation and to facilitate awareness of internal cues related to desire, motivation, and individual responses to stress.

Researchers will compare usual prenatal care plus TPI versus usual prenatal care plus prenatal education to see if TPI reduces psychological (e.g., depression, anxiety, and perceived stress), and socio-emotional (e.g., mood, resilience, social support), and prenatal health behaviors.

DETAILED DESCRIPTION:
The goal of this research to reduce the impact of maternal adverse childhood experiences (ACEs) on perinatal mental and psychosocial health by providing the necessary tools for the development of healthy coping practices. The purpose of this proposal is to conduct Phase II preliminary testing of an individually randomized pilot trial (N=40) examining feasibility, acceptability, and compare initial estimates of the effects of the primary outcome of depression and secondary outcomes of psychological (e.g., stress and anxiety) and socio-emotional (e.g., mood, resilience, social support) functioning and prenatal health behaviors of those allocated to either a trauma-informed prenatal intervention (TPI) (n=15) or the control group, e.g., prenatal education arm, (n=15). Forty adult, pregnant women receiving prenatal care at one large Federally Qualified Health Center will be enrolled between 10-24 weeks gestation. TPI participants will receive four weekly (30-60 minute) individual online sessions of motivational interviewing to facilitate behavior change and mental wellness skills to promote self-regulation. Control group participants will receive four weekly (30-60 minutes) individual online sessions of prenatal education. Patient-reported outcome measures will be interview-administered at baseline, 4- and 12-weeks post-randomization, and 6-weeks postpartum. A trauma-informed approach within prenatal care services may help reduce maternal distress and its consequences, and, subsequently, lessen the risk for the negative impact of ACEs on maternal and child health. Findings from this study will inform a larger efficacy trial of TPI to improve perinatal mental health among pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* receiving prenatal care at University of Illinois Health & Hospital System
* age >/= 18 years
* English-speaking
* 10-24 weeks gestation
* able to attend four sessions
* owner of a smart phone and access to internet

Exclusion Criteria: inability to reliably or safely participate in the study due to self-reported serious or persistent mental health disorder (e.g., schizophrenia or bipolar disorder), which could also interfere with study adherence.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant people
Enrollment: 40 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Edinburgh Postnatal Depression Scale at 2-months post-intervention | 6-weeks postnatal
  The Edinburgh Postnatal Depression Scale (range: 0-30) is a 10-item scale is a pregnancy and/or postpartum depression screen that assesses different emotions in the past seven days in which a higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder Scale at 2-months post-intervention | 6-weeks postnatal
  Generalized Anxiety Disorder Scale (range: 0-21) is a 7-item scale that assesses the frequency of excessive, uncontrollable worry in the past two-weeks in which a higher score indicates a worse outcome regarding life events or activities in which a higher score signifies a worse outcome.
Change in Perceived Stress Scale at 2-months post-intervention | 6-weeks postnatal
  The Perceived Stress Scale (range: 0-40) is a 10-item scale that assesses the frequency of stressful thoughts and feelings in the last one month in which a higher score indicates a worse outcome.
Change in Behavioral Activation Scale at 2-months post-intervention | 6-weeks postnatal
  The Behavioral Activation Scale (range: 0-54) is a 9-item scale that assesses avoidance or engagement in goal-directed activity and pleasant behaviors during the past one week in which a higher score indicates a better outcome.
Negative Mood Regulation Short Form Scale at 2-months post-intervention | 6-weeks postnatal
  The Negative Mood Regulation Scale (range: 15-75) is a 15-item scale that assesses the capacity for calming and soothing emotions when one is upset in which a higher score indicates a better outcome.
Connor Davidson Resilience Scale at 2-months post-intervention | 6-weeks postpartum
  The 10-item CD-RS assesses resilience over the last month. Responses are scored on a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all the time), with high scores representing greater ability to bounce back from adversity.
Prenatal Health Behaviors at 2-months post-intervention | 6-weeks postnatal
  The Prenatal Health Behaviors Scale (range: 0-96) is a 24-item scale that assesses the frequency of the use of prenatal health behaviors, including smoking, alcohol, drugs, food, vitamins, physical activity, sleep, etc in which a higher score signifies a worse outcome.
Multidimensional Scale of Perceived Social Support at 2-months post-intervention | 6-weeks postpartum
  The 12-item MSPSS assesses social support from family, friends, and a significant other. Responses are scored on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree), with high scores representing greater perceived social support.

OTHER OUTCOMES:
Prenatal Distress at 2-months post-intervention | 2-months post-intervention
  The Prenatal Distress Scale (range: 0-35) is an 18-item scale that assesses the things that are worrisome or bothersome about their pregnancy in which a higher score indicates a worse outcome.
Treatment Acceptability and Preferences Scale at post-intervention | 4-weeks post-randomization
  The Treatment Acceptability and Preferences Scale (range: 0-36) is a 9-item scale that evaluates the effectiveness, acceptability, and suitability of the intervention in which a higher score indicates a better outcome.
Expanded Adverse Childhood Experiences at baseline | Baseline
  The Expanded Adverse Childhood Experiences survey (range: 0-21) is a 21-item questionnaire that assesses childhood adversity prior to age 18 years in which a higher score indicates a worse outcome.
Benevolent Childhood Experiences at baseline | Baseline
  The Benevolent Childhood Experiences survey (range: 0-10) is a 10-item questionnaire that assesses positive childhood experiences during your first 18 years of life in which a higher score indicates a worse outcome.
Everyday Discrimination Scale at baseline | Baseline
  The Everyday Discrimination Scale (range: 0-50) assesses the frequency of negative experiences as a result of one's race, ethnicity, or skin color in which a higher score indicates a worse outcome. The EDS was developed as a subjective measure to capture self-reported frequency of routine, relatively subtle discriminatory experiences in everyday social situations. Responses are typically coded on a 6-point Likert scale ranging from 'never' to 'almost everyday'.
Social Determinants of Health Assessment Tool at baseline | Baseline
  The Social Determinants of Health Assessment Tool is a 10-item survey (0-10) that helps to identify health-related social needs (e.g., food, housing/utilities, transportation, and personal safety.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Goldstein, PhD, MFT, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Health & Hospital System, Chicago, Illinois, United States

REFERENCES:
- [Derived] Goldstein E, Keita M, Koomson C, Tintle N, Adlam K, Farah E, Koenig MD. A Pilot Randomized Controlled Trial of a Multimodal Wellness Intervention for Perinatal Mental Health. J Midwifery Womens Health. 2025 May-Jun;70(3):442-451. doi: 10.1111/jmwh.13754. Epub 2025 Apr 10. PMID 40207735
- [Derived] Itani MS, Shankar M, Goldstein E. Exploring trauma-informed prenatal care preferences through diverse pregnant voices. BMC Health Serv Res. 2025 Mar 27;25(1):452. doi: 10.1186/s12913-025-12519-w. PMID 40148939